CLINICAL TRIAL: NCT04420182
Title: COVID-19 Virtual Care at Home
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's (Other)
Collaborators: Cardiac Arrhythmia Network of Canada (Other)
Responsible Party: Principal Investigator, Anthony Tang, Principal Investigator, London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CTO 3210
Record Dates: First submitted 2020-05-29; First posted 2020-06-09 (Actual); Last update posted 2022-04-07 (Actual); Status verified 2022-04

CONDITIONS: Covid-19
Keywords: COVID-19; SARS-CoV-2; VIRTUES; Virtual Care Management; Virtual Care; Patient Satisfaction; Anxiety; Emergency Visits; Oxygen Saturation; Quality of Life
MeSH Terms: conditions — COVID-19; Patient Satisfaction; Anxiety Disorders

STUDY DESIGN:
Intervention Model Description: Prospective non-randomized cohort study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- COVID-19 Virtual Care at Home (Other): VIRTUES COVID-19 Care at Home Platform
  The components of the platform will include:
  1. Vital sign monitoring, including O2 saturation with a home-based pulse oximeter, temperature and respiratory rate performed three times per day (a notification to do this will be sent from the app), with the option of doing assessments more frequently if needed. Study patients will be provided monitoring devices to collect this data.
  2. Symptom logs will be entered by the patients.
  3. Feedback to the patient by the local COVID-19 care team for any action:
     1. Two-way communication between the patient and the COVID-19 care team
     2. Ability for team members to see all prior notes in order to have continuity of care
     3. Reports of these interactions are transmitted to the patient's health record
  4. Current information on COVID-19 as per the Public Health Agency of Canada
  Interventions: Other: Virtual Care at Home

INTERVENTIONS:
Other: Virtual Care at Home — Participants will have access to the VIRTUES platform for COVID-19 Virtual Care at Home

SUMMARY:
This multicentre prospective cohort trial is designed to demonstrate effectiveness and efficiency of a virtual care model for the management of COVID-19 patients isolating at home. The investigators have reoriented existing technology and networks for this research project. The investigators are amplifying our existing virtual care platform VIRTUES, combining it with home monitoring of COVID-19 patients, to provide real-time evidence, harmonize data collection, and share data provincially to mitigate the impact of the rapid spread of the virus. The study will facilitate early detection of complications associated with the disease, treatment and management of COVID-19 patients at home. The research will be conducted provincially in Ontario.

This initiative will provide evidence to inform clinical and health system management and public health response to COVID-19 patients isolating at home.

ELIGIBILITY:
Inclusion Criteria:

* All COVID-19 positive patients of age 18 or above
* Participant must communicate in English or French language
* An email address and account

Exclusion Criteria:

* Unable or unwilling to provide informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 817 (Actual)
Dates: Start 2020-08-17 (Actual); Primary Completion 2022-02-04 (Actual); Study Completion 2022-02-04 (Actual)

PRIMARY OUTCOMES:
14 Day Patient Satisfaction Questionnaire | 14 days
  The primary outcome measure is patient satisfaction as measured from a patient satisfaction questionnaire at 14 days.

SECONDARY OUTCOMES:
Emergency Department Visits | 14 days
  The secondary outcome measures will include the number of patients that require an Emergency Department visits during the observation period of 14 days.
14 Day EQ-5D-5L Scores | 14 days
  The secondary outcome measures will include the health status measures of the EuroQuality of Life Five Dimensions (EQ-5D-5L) at 14 days. Scoring is Level 1 to 5 for each dimension; higher scores meaning worse health status.

CONTACTS AND LOCATIONS:
Locations (5):
- Canada (5):
  - St. Mary's General Hospital, Kitchener, Ontario
  - London Health Sciences Centre, London, Ontario
  - Ottawa Heart Research Institute, Ottawa, Ontario
  - Niagara Health, St. Catharines, Ontario
  - St. Joseph's Health Centre, Toronto, Ontario